CLINICAL TRIAL: NCT02719353
Title: A Dispensing Clinical Trial of Comfilcon A Extended Range Multifocal Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV-16-02
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- comfilcon A Extended Range test lens (Experimental): Subjects will be randomized to wear either the test or control pair of lens, then cross over to the alternate pair.
  Interventions: Device: comfilcon A Extended Range test lens; Device: comfilcon A control lens
- comfilcon A control lens (Active Comparator): Subjects will be randomized to wear either the test or control pair of lens, then cross over to the alternate pair.
  Interventions: Device: comfilcon A Extended Range test lens; Device: comfilcon A control lens

INTERVENTIONS:
Device: comfilcon A Extended Range test lens — contact lens
Device: comfilcon A control lens — contact lens

SUMMARY:
The aim of this study is to validate the clinical of comfilcon A extended range high add center near (CN) multifocal lenses in existing contact lens wearers against the current comfilcon A high add multifocal lenses.

DETAILED DESCRIPTION:
This study is a 13-subject, randomized, prospective, single site, daily wear, single-masked (to the subject), bilateral, 4-day cross-over, dispensing study comparing the comfilcon A extended range multifocal test lens against the comfilcon A multifocal control lens.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Has had a self-reported oculo-visual examination in the last two years
* Is 50 years of age or greater and has full legal capacity to volunteer
* Is able to read and understand the informed consent
* Is willing and able to follow instructions and maintain the appointment schedule
* Has a spherical distance contact lens prescription between -1.00 and -5.00D (Diopters) (inclusive)
* Near Add Power requirement of +2.25D or greater
* Has spectacle cylinder 0.75 D in both eyes
* Has normal binocularity (no amblyopia, no strabismus, no habitually uncorrected anisometropia ≥ 2.00D)
* Has monocular best-corrected distance visual acuity of 20/30 or better in each eye
* Has clear corneas and no active ocular disease
* Has not worn gas permeable contact lenses for 1 month prior to the study

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before
* Has any systemic disease affecting ocular health
* Is using any systemic or topical medications that will affect ocular health
* Has any ocular pathology or abnormality that would affect the wearing of contact lenses
* Is aphakic (i.e. missing their natural lens inside their eye)
* Has uncorrected anisometropia (i.e. difference in the prescription between the eyes) of ≥2.00 D
* Has undergone corneal refractive surgery
* Is participating in any other type of eye related clinical or research study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete S Kollbaum, O.D., Principal Investigator — Indiana University
Locations (1):
- CORL, Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Lens Then Control Lens: Subjects will be randomized to wear the test contact lenses then control contact lenses bilaterally for four days in the cross-over study.
  comfilcon A Extended Range test lens: contact lenses comfilcon A control lens: contact lenses
- Control Lens Then Test Lens: Subjects will be randomized to wear the control contact lenses then test contact lenses bilaterally for four days in the cross-over study.
  comfilcon A control lens: contact lenses comfilcon A Extended Range test lens: contact lenses
Period: First Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Second Intervention
Arm/Group | Test Lens Then Control Lens | Control Lens Then Test Lens
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects will be randomized to wear the test contact lenses or control contact lenses first as per the randomization table bilaterally for four days then cross-over to alternated pair lenses.
  comfilcon A Extended Range test lens: contact lenses comfilcon A control lens: contact lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was measured at distance, intermediate and near conditions for test and control lens was assessed by LogMAR.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Comfilcon A Extended Range Test Lens: Subjects will be randomized to wear the test contact lenses bilaterally for four days in this cross-over study.
  comfilcon A Extended Range test lens: contact lens
- Comfilcon A Control Lens: Subjects will be randomized to wear the control contact lenses bilaterally for four days in this cross-over study.
  comfilcon A control lens: contact lens
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
LogMAR
  Distance | -0.01 (0.09) | -0.07 (0.10)
  Intermediate | -0.15 (0.16) | -0.13 (0.10)
  Near | -0.02 (0.09) | 0.01 (0.07)

2. Primary Outcome: Visual Performance
Description: Subjective assessment of visual performance for test and control lens is assessed on a scale 0-100, 0=extremely poor vision all of the time and cannot function, 100= excellent vision all of the time).
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale
  Distance | 72 (19) | 77 (20)
  Intermediate | 85 (17) | 88 (13)
  Near | 79 (23) | 80 (16)

3. Secondary Outcome: Subjective Ratings for Comfort
Description: Subjective ratings for comfort was assessed for test and control lens on a Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 96 (8) | 91 (6)

4. Secondary Outcome: Subjective Ratings for Comfort
Description: as for outcome 3
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 87 (21) | 89 (17)

5. Secondary Outcome: Subjective Ratings for Dryness
Description: Subjective ratings for dryness was assessed for test and control lens on a scale 0-100, 0=cannot be worn, extremely dry, 100=no dryness experienced at any time).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 94 (9) | 94 (7)

6. Secondary Outcome: Subjective Ratings for Dryness
Description: as for outcome 5
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 83 (23) | 88 (14)

7. Secondary Outcome: Lens Handling
Description: Subjective ratings for handling (ease of insertion and removal) was assessed for test and control lens on a scale 0-100, 0=very difficult to handle, 100=easy to handle).
Time Frame: 4 Days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 89 (25) | 95 (9)

8. Secondary Outcome: Average Daily Wearing Time
Description: Average daily wearing time for test and control lens is assessed in hours.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
Hours/day | 10 (2) | 9 (3)

9. Secondary Outcome: Lens Fit
Description: Lens fit acceptance (general fit characteristics) is assessed for test and control lens on a 0-4 grading system in 0.25 steps where 0 represented very poor fit.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 3.3 (0.4) | 3.3 (0.3)

10. Secondary Outcome: Bulbar Hyperemia
Description: Bulbar hyperemia was assessed on a scale of 0-4 and was used in 0.50 steps, with 0 indicating no hyperemia and 4 indicating severe hyperemia.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 0.88 (0.44) | 0.89 (0.42)

11. Secondary Outcome: Limbal Hyperemia
Description: Limbal hyperemia was assessed on a scale of 0-4 and was used in 0.50 steps, with 0 indicating no hyperemia and 4 indicating severe hyperemia.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 0.13 (0.26) | 0.18 (0.28)

12. Secondary Outcome: Subjective Satisfaction
Description: Subjective satisfaction for test and control lens was assessed on a scale 0-100, 0=extremely dissatisfied, 100=very satisfied)
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 13 | 13
units on a scale | 71 (23) | 74 (19)

13. Secondary Outcome: Subjective Preference for Near Vision
Description: Subjective preference for near vision for test and control contact lenses. comfort, vision, handling, satisfaction.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Subjects were randomized to wear test lens or control contact lenses bilaterally for four days in this cross-over study.
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Test | 4
  No Preference | 4
  Control | 5

14. Secondary Outcome: Subjective Preference for Distance Vision
Description: Subjective preference for distance vision for test and control contact lenses.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Test | 3
  No Preference | 2
  Control | 8

15. Secondary Outcome: Subjective Preference for Intermediate Vision
Description: Subjective preference for intermediate vision for test and control contact lenses.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Test | 3
  No Preference | 4
  Control | 6

16. Secondary Outcome: Subjective Preference for Overall Vision
Description: Subjective preference for overall vision for test and control contact lenses.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Test | 3
  No Preference | 1
  Control | 9

17. Secondary Outcome: Subjective Preference for Comfort
Description: Subjective preference for comfort for test and control contact lenses.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Test | 4
  No Preference | 3
  Control | 6

18. Secondary Outcome: Subjective Overall Lens Preference
Description: Subjective overall lens preference for test and control contact lenses.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Test | 4
  No Preference | 0
  Control | 9

ADVERSE EVENTS:
Time Frame: From dispense up to four days on each pair of contact lenses.
Arm/Group | Comfilcon A Extended Range Test Lens | Comfilcon A Control Lens
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No